A Randomized Controlled Trial of Acetaminophen and Ibuprofen Versus Acetaminophen and Oxycodone for Postoperative Pain Control in Operative Pediatric Supracondylar Humerus Fracture

NCT03759028

Unique Protocol ID# 18-001158

Date of Document: 11/14/2018

## UNIVERSITY OF CALIFORNIA LOS ANGELES

## ASSENT TO PARTICIPATE IN RESEARCH

A Randomized Controlled Trial of Acetaminophen and Ibuprofen Versus Acetaminophen and Oxycodone for Postoperative Pain Control in Operative Pediatric Supracondylar Humerus Fractures

- 1. My name is Dr. Rachel Thompson/Dr. Mauricio Silva.
- 2. We are asking you to take part in a research study because we are trying to learn more about pain control after elbow surgery
- 3. If you agree to be in this study you will be asked about your pain levels at various time points after surgery.
- 4. You may experience that the pain medication may not work well; in that case, you can have your parents ask for another medication that the pharmacy will give you
- 5. You may potentially avoid strong medication which can make you feel sick
- 6. Please talk this over with your parents before you decide whether or not to participate. We will also ask your parents to give their permission for you to take part in this study. But even if your parents say "yes" you can still decide not to do this.
- 7. If you don't want to be in this study, you don't have to participate. Remember, being in this study is up to you and no one will be upset if you don't want to participate or even if you change your mind later and want to stop.
- 8. You can ask any questions that you have about the study. If you have a question later that you didn't think of now, you can call me at 213.742.1369 or ask me next time. You may call me at any time to ask questions about your disease or treatment.
- 9. Signing your name at the bottom means that you agree to be in this study. Your doctors will continue to treat you whether or not you participate in this study. You and your parents will be given a copy of this form after you have signed it.

| Name of Subject | Date |
|-----------------|------|